CLINICAL TRIAL: NCT02257281
Title: Chung Shan Medical University Hospital Institutional Review Board
Brief Title: The Effect of Therapeutic Ultrasound on Soft Tissue: An Experimentally-induced Skin Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, GCRC, Chung Shan Medical University, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS14008
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Inflammation
Keywords: Sodium lauryl sulfate; Skin irritants; inflammation; therapeutic ultrasound
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Therapeutic Ultrasound (Experimental): The three inflammatory forearm spots on the same side induce by the experimentally skin model(1%, 0.5%, 0% SLS) treat with active therapeutic ultrasound .
  Interventions: Device: Active Therapeutic Ultrasound
- Non-active Therapeutic Ultrasound (Placebo Comparator): The contralateral three inflammatory forearm spots induce by the experimentally skin model(1%, 0.5%, 0% SLS) treat with non-active therapeutic ultrasound .
  Interventions: Device: Non-active Therapeutic Ultrasound

INTERVENTIONS:
Device: Active Therapeutic Ultrasound — For Experimental Arm: The pulsed therapeutic ultrasound was applied each spot for several days.
  Arms: Active Therapeutic Ultrasound
Device: Non-active Therapeutic Ultrasound — For Placebo group: The non-active therapeutic ultrasound was applied each spot for several days.
  Arms: Non-active Therapeutic Ultrasound

SUMMARY:
The purposes of study are to investigate the effect of therapeutic ultrasound for the inflammatory skin repair and whether the tissue repair under ultrasound treament is depend on different inflammatory level.

DETAILED DESCRIPTION:
Therapeutic ultrasound for soft tissue repair has been used in clinical during the past decades. In some recent systematic review, the evidence of clinical trials were insufficiency. We assumed the reaserch biasin clinical trials may be due to the different inflammatory level of soft tissue under the similar ultrasound intensity. Our purpose of study is to investigate the effect of therapeutic ultrasound for the inflammatory skin repair and whether the tissue repair under ultrasound treament is depend on different inflammatory level.

ELIGIBILITY:
Inclusion Criteria:

1. asia healthy subjects
2. aged 20-45 years

Exclusion Criteria:

1. disadvantaged groups
2. systemic disease, such as DM, cancer, autoimmune disorder
3. hyperhidrosis or hypothyroidism
4. a past history of dermatitis
5. active infective or inflammatory cutaneous disease
6. smoking or drinking
7. take medicine, over sun exposure, exercise or menstruation during experimental period
8. contraindication of therapeutic ultrasound

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
skin blood flow | 2 weeks

SECONDARY OUTCOMES:
skin temperature | 2 weeks
skin water content | 2 weeks
Tactile pain threshold | 2 weeks
erythema index | 2 weeks
skin thickness | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peir Renn Wang, MD, Principal Investigator — Department of rehabilitation